CLINICAL TRIAL: NCT04374656
Title: Prevalence of SARS-CoV-2 in Conjunctival Swab Samples Among Patients Presenting With Conjunctivitis to the Ophthalmology Clinics During the COVID-19 Pandemic
Brief Title: Prevalence of SARS-CoV-2 in Conjunctival Swab Samples Among Patients With Conjunctivitis During the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00249598
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Conjunctivitis; SARS-CoV-2; COVID-19; Ocular Infection, Viral; Ocular Inflammation
Keywords: conjunctivitis; SARS-CoV-2; COVID-19; Ocular Infection; viral conjunctivitis; ocular inflammation; conjunctival swab; PCR
MeSH Terms: conditions — Conjunctivitis; COVID-19; Eye Infections, Viral; Eye Infections; Conjunctivitis, Viral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Conjunctival, nasal, and nasopharyngeal swabs will be taken for PCR testing and next-generation sequencing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) is a newly identified, highly contagious RNA virus causing respiratory infectious disease, Coronavirus Disease 2019 (COVID-19). Conjunctivitis has been reported as a rare finding of the disease, and preliminary studies showed that the virus RNA could be detected in ocular secretions using polymerase chain reaction (PCR) assays when conjunctivitis present. This study aims to estimate the proportion of SARS-CoV-2 associated conjunctivitis among patients with suspected viral conjunctivitis presented to the ophthalmology clinics of Wilmer Eye Institute during the COVID-19 pandemic. The investigators also aim to identify whether SARS-CoV-2 associated conjunctivitis is an isolated finding or an early sign of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older
* Willingness to participate
* Presents with red eye complaint

Exclusion Criteria:

* Adults lacking capacity to consent
* Adults with special needs due to physical, medical, developmental or cognitive conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients present or are referred to the ophthalmology clinic due to red eye complaints, suspected viral conjunctivitis, or keratoconjunctivitis will be consecutively approached and recruited if they show a willingness to participate.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2020-05-18 (Actual); Primary Completion 2024-05-29 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Proportion of conjunctival samples tested positive for SARS-CoV-2 | 1 year
  Number of conjunctival samples with positive PCR divided by the total number of conjunctival samples

SECONDARY OUTCOMES:
Proportion of nasal samples tested positive for SARS-CoV-2 among patients with positive conjunctival samples | 1 year
  Number of nasal samples with positive PCR divided by the number of conjunctival samples with positive PCR
Proportion of nasopharyngeal samples tested positive for SARS-CoV-2 among patients with positive conjunctival samples | 1 year
  Number of nasopharyngeal samples with positive PCR divided by the number of conjunctival samples with positive PCR
Rate of development of COVID-19 in the study patient population | 1 year
  Number of patients developed COVID-19 divided by the number of the study population
Positive conjunctival sample rate in patient developed COVID-19 | 1 year
  Number of conjunctival samples with positive PCR divided by the number of patients developed COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Sezen Karakus, MD, Principal Investigator — Wilmer Eye Institute at Johns Hopkins University
Locations (1):
- Wilmer Eye Institute, Baltimore, Maryland, United States